CLINICAL TRIAL: NCT05332561
Title: Genomics Guided Targeted Post-neoadjuvant Therapy in Patients With Early Breast Cancer - a Multicenter, Open-label, Umbrella Phase-II Study - COGNITION-GUIDE
Brief Title: Genomics Guided Targeted Post-neoadjuvant Therapy in Patients With Early Breast Cancer (COGNITION-GUIDE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DKFZ-2019-008; 2020-002606-22 (EudraCT Number); 01EK2202A (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF)); 2024-514022-23-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-22; First posted 2022-04-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Early-stage Breast Cancer
Keywords: Breast Cancer; Post-neoadjuvant therapy; genomics-guided; molecular diagnostic; targeted therapy; high risk
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Injections; inavolisib; ipatasertib; olaparib; sacituzumab govitecan; Trastuzumab; pertuzumab

STUDY DESIGN:
Intervention Model Description: Umbrella
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Arm 1 Atezolizumab (Immune Evasion) (Experimental): Atezolizumab Dosage: 1200 mg, intravenous, on d1, q21d
  Interventions: Drug: Atezolizumab 1200 mg in 20 ML Injection
- Arm 2 Inavolisib (PI3K) (Experimental): Inavolisib Dosage: 9 mg, oral, on d1-d28, q28d
  Interventions: Drug: Inavolisib
- Arm 3 Ipatasertib (AKT) (Experimental): Ipatasertib Dosage: 400 mg, oral, on d1-d21, q28d
  Interventions: Drug: Ipatasertib
- Arm 4 Olaparib (PARP, DNA-Repair) (Experimental): Olaparib Dosage: 300 mg, oral, bid d1-d28, q28d
  Interventions: Drug: Olaparib
- Arm 5 Sacituzumab Govitecan (TROP-2) (Experimental): Sacituzumab Govitecan Dosage: 10 mg/kg BW, intravenous, on d1 and d8, q21d
  Interventions: Drug: Sacituzumab govitecan
- Arm 6 Trastuzumab/Pertuzumab (ERBBB) (Experimental): Trastuzumab/Pertuzumab Administration: subcutaneous; Initial dose: Trastuzumab 600 mg, Pertuzumab 1200 mg, 30 000 units hyaluronidase; Maintainance dose: Trastuzumab 600 mg, Pertuzumab 600 mg, 20 000 units hyaluronidase; Frequency: on d1, q21d
  Interventions: Drug: Trastuzumab/pertuzumab
- Arm 7 Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Atezolizumab 1200 mg in 20 ML Injection — Arm 1
  Other Names: Tecentriq
  Arms: Arm 1 Atezolizumab (Immune Evasion)
Drug: Inavolisib — Arm 2
  Arms: Arm 2 Inavolisib (PI3K)
Drug: Ipatasertib — Arm 3
  Arms: Arm 3 Ipatasertib (AKT)
Drug: Olaparib — Arm 4
  Other Names: Lynparza
  Arms: Arm 4 Olaparib (PARP, DNA-Repair)
Drug: Sacituzumab govitecan — Arm 5
  Other Names: Trodelvy
  Arms: Arm 5 Sacituzumab Govitecan (TROP-2)
Drug: Trastuzumab/pertuzumab — Arm 6
  Other Names: Phesgo
  Arms: Arm 6 Trastuzumab/Pertuzumab (ERBBB)

SUMMARY:
In early breast cancer (eBC), pathological complete response (pCR) after neoadjuvant therapy acts as surrogate marker for metastasis and overall survival. Therapy intensification by adding an adjuvant therapy line (post-neoadjuvant treatment) substantially lowers the risk of relapse in high-risk breast cancer patients with residual disease after neoadjuvant treatment (non-pCR). While this approach was exemplified in two phase III trials without biomarker-stratification (CREATE-X, KATHERINE), even higher efficiency might be achieved by individualized genomic-guided post-neoadjuvant therapies.

Within the seven-arm umbrella phase-II clinical trial COGNITION-GUIDE, we aim to deliver molecularly-tailored cancer care by implementing an additional response- and genomics-guided post-neoadjuvant therapy after finishing the guideline-compliant post-neoadjuvant treatment in high-risk breast cancer patients with residual cancer burden after neoadjuvant therapy to reduce the substantial risk of local and distant relapse.

The trial evaluates not a single drug but rather a general strategy of precision oncology in the curative setting and provides the basis for future confirmatory biomarker-driven trials.

Allocation to the therapy-arms is conducted by in depth molecular characterization of tumors within the COGNITION registry program.

The study aims to show an overall benefit of the precision medicine approach in high-risk eBC patients and to allow for secondary exploratory evaluation of each study-arm.

The primary endpoint of the study is invasive Disease-Free Survival (IDFS) after 4 years measured from surgery to local or distant relapse or death. The sample size of the entire trial is 240 eligible patients.

DETAILED DESCRIPTION:
In early breast cancer (eBC), pathological complete response (pCR) after neoadjuvant therapy acts as surrogate marker for metastasis and overall survival.

Therapy intensification by adding an adjuvant therapy line (post-neoadjuvant treatment) substantially lowers the risk of relapse in high-risk breast cancer patients with residual disease after neoadjuvant treatment (non-pCR).

While this approach was exemplified in two phase III trials without biomarker-stratification (CREATE-X, KATHERINE), even higher efficiency might be achieved by individualized genomic-guided post-neoadjuvant therapies.

To date, prospective whole genomic and transcriptomic sequencing in the framework of precision oncology concepts is predominantly conducted in advanced-stage cancer, limiting the overall benefit mainly to prolongation of progression-free survival rather than cure.

In contrast, the implementation of precision oncology in an early disease stage may empower targeted intervention based on high throughput sequencing at a time point with low tumor burden and limited clonal complexity, harbouring the prospect to substantially improve cure rates by prohibition of incurable metastasis.

Whole-genome (WGS), whole exome (WES), gene panel and transcriptome sequencing in the molecular diagnostic registry platform COGNITION (neoadjuvant-treated eBC patients) revealed relevant diagnostic information on molecular-druggable alterations in a substantial proportion of patients in different molecular pathways (e.g. phosphatidylinositol 3-kinase (PI3K)/ serine/threonine kinase (AKT), Mitogen-activated protein kinase (MAPK), apoptosis, DNA-repair, immune escape etc.).

Within the seven-arm umbrella phase-II clinical trial COGNITION-GUIDE, we aim to deliver molecularly-tailored cancer care by implementing an additional response- and genomics-guided post-neoadjuvant therapy after finishing the guideline-compliant post-neoadjuvant treatment in high-risk breast cancer patients with residual cancer burden after neoadjuvant therapy to reduce the substantial risk of local and distant relapse.

The trial evaluates not a single drug but rather a general strategy of precision oncology in the curative setting and provides the basis for future confirmatory biomarker-driven trials.

Eligible patients are identified considering pCR-status and clinical stage estrogen receptor status grade (CPS-EG)-score following surgery after neoadjuvant therapy.

Allocation to the therapy-arms is conducted by in depth molecular characterization of tumors within the COGNITION registry program.

Recruitment of adequate patient numbers in well-defined molecular subgroups is achieved in a multicenter approach.

The study aims to show an overall benefit of the precision medicine approach in high-risk eBC patients and to allow for secondary exploratory evaluation of each study-arm.

The primary endpoint of the study is invasive Disease-Free Survival (IDFS) after 4 years measured from surgery to local or distant relapse or death.

The sample size of the entire trial is 240 eligible patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Female and male patients with non-metastatic early (stage I-III) breast cancer aged ≥ 18 years
3. Conducted neoadjuvant chemotherapy and surgery as well as conducted standard post-neoadjuvant treatment +/- radiotherapy (standard according to German guidelines except Abemaciclib and Olaparib)
4. For patients with initially triple negative (TNBC) or HER2-positive breast cancer:

   • Non-pCR defined as other than ypT0/is ypN0
5. For patients with initially hormone receptor positive and HER2-negative breast cancer: Non-pCR and CPS-EG score

   * ≥ 3 and ypN0, or
   * ≥ 2 and ypN+
6. ECOG Performance Status ≤ 1
7. Acute effects of any prior therapy resolved to baseline severity or National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0) Grade ≤ 1 except for adverse effects not constituting a safety risk by investigator judgement
8. Postmenopausal or evidence of non-childbearing status. For women of childbearing potential negative urine pregnancy test at post-operative screening and baseline as well as highly effective forms of contraception have to be in place thereafter

   * Evidence of childbearing potential is defined as fertile, following menarche and until becoming post-menopausal unless permanently sterile
   * Postmenopausal or evidence of non-childbearing status is defined as:

     * Amenorrhea for 1 year or more without an alternative medical cause following cessation of exogenous hormonal treatments plus follicle stimulating hormone (FSH) levels in the postmenopausal range in women not using hormonal contraception or hormonal replacement therapy
     * Chemotherapy-induced menopause
     * Surgical sterilisation (bilateral oophorectomy, bilateral salpingectomy, total hysterectomy or tubal ligation at least 6 weeks before IMP treatment)
     * Female patients with age ≥ 60 years
   * A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy
9. Female patients of childbearing potential and male patients with partners of childbearing potential who are sexually active must agree to the use of two forms of contraception in combination (male condom and one highly effective method). These should be started immediately after signing the informed consent form and continued throughout the period of study treatment plus a substance-depending time period (see respective sub-protocol) for female patients and a substance-depending time period for male patients. Details on contraception and pregnancy testing for male and female patients (and if indicated their partners) under IMP treatment are described within the respective sub-protocol
10. Ability of patient to understand and comply with the protocol for the duration of the study, including treatment and scheduled visits and examinations
11. Adequate bone marrow, renal, and hepatic function defined by laboratory tests*

The biomarker-guided eligibility for the respective study arm is evaluated and determined exclusively by the NCT molecular tumor board on the basis of results of the COGNITION molecular diagnostic registry platform. Biomarkers that allow inclusion in the respective arm are:

* Arm 1 (Atezolizumab, Immune Evasion ): PD-L1 positivity measure by IHC (≥1% on immune cells within the tumor), MSI-high status (validated by PCR), TMB-H (≥10mut/MB), CD274 amplification
* Arm 2 (Inavolisib, PI3K): Known/reported oncogenic mutation in PIK3Ca
* Arm 3 (Ipatasertib, AKT): Aberrations predicting increased PI3K-AKT pathway activity except PI3K-mutations, HR positive histology
* Arm 4 (Olaparib, PARP, DNA-Repair): Inactivating somatic or germline BRCA1/2 mutation including homozygous deletions, Inactivating germline PALB2 mutations
* Arm 5 (Sacituzumab Govitecan, TROP-2): Trop-2-overexpression (with IHC and except known/reported homozygous polymorphism in UGT1A1*28)
* Arm 6 (Trastuzumab / Pertuzumab, ERBBB): HER2 exon-20 insertion, Activating HER2-mutation

Exclusion Criteria:

1. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1 grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥ 5 year
2. Concurrent severe, uncontrolled systemic disease that would place patient at undue risk or interfere with planned treatment
3. Concurrent participation or previous treatment within 30 days in another interventional clinical trial
4. Persistent toxicity (≥ Grade 2 according to NCI CTCAE v5.0 caused by previous cancer therapy, excluding alopecia
5. Clinical signs of active infection (> Grade 2 according NCI CTCAE v5.0)
6. History of or newly diagnosed human immunodeficiency virus (HIV) infection and immunocompromised patients
7. Active Hepatitis A virus infection
8. Active hepatitis B virus (HBV) infection, defined as having a positive hepatitis B surface antigen (HBsAg) test. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening, are eligible for the study if active HBV infection is ruled out on the basis of HBV DNA viral load per local guidelines
9. Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test at screening confirmed by a polymerase chain reaction (PCR) positive for HCV RNA
10. Dementia or significant impairment of cognitive state
11. Epilepsy requiring pharmacologic treatment
12. Pregnancy and breast feeding
13. Inability to take oral medication and gastrointestinal disorders likely to interfere with absorption of study medication
14. Major surgery (any invasive operative procedure in which a more extensive resection is performed, e.g. a body cavity is entered, organs are removed, or normal anatomy is altered) within four weeks before screening and baseline excluding breast-tumor resection after neoadjuvant chemotherapy. Patients must have recovered from any effects of any major surgery
15. Systemic chemotherapy or radiotherapy within four weeks or a longer period depending on the characteristics of the agents used
16. Heart failure classified as New York Heart Association (NYHA) II/III/IV
17. Severe obstructive or restrictive ventilation disorder
18. Patients with clinically active tuberculosis
19. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug
20. Is taking or requiring the continued use of any of the prohibited concomitant medications listed in the respective subprotocols at baseline
21. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder or non-malignant systemic disease. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression or, superior vena cava syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (IDFS) as defined by Hudis et al in the entire study population four years after surgery | Four years after surgery
  Primary objective is to improve clinical outcome in early high-risk breast cancer by biomarker-guided post-neoadjuvant therapy (systemic treatment in the adjuvant setting following neoadjuvant therapy, surgery and post-neoadjuvant standard therapy)

SECONDARY OUTCOMES:
Invasive Disease-free Survival (IDFS) as defined by Hudis et al | Four years after surgery
  in each study arm separately
Distant Disease-free Survival (DDFS) as defined by Hudis et al | Four years after surgery
  in each study arm separately and overall
Overall Survival | When the last patient has completed four years after surgery
  in each study arm separately and overall
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | Through treatment period of the study, an average of 1 year
  in each study arm separately and overall

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schneeweiss, Prof. Dr., Principal Investigator — National Center for Tumor Diseases (NCT)
Locations (9):
- Germany (9):
  - National Center for Tumor Diseases, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Ulm, Ulm, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Carl-Gustav-Carus, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen, Essen

DOCUMENTS (1):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT05332561/Prot_000.pdf